CLINICAL TRIAL: NCT04760639
Title: Breath Test Feasibility Trial for COVID-19 Infection Diagnosis
Brief Title: COVID Breath Test - Ancon
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Gerard Silvestri, MD, Professor of Medicine, Medical University of South Carolina
Other Study IDs: Pro00102970
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test group: Participants who have a positive Covid-19 Test or negative Covid-19 test who provide a breath sample.
  Interventions: Diagnostic Test: Breath test

INTERVENTIONS:
Diagnostic Test: Breath test — Participants provide a breath sample

SUMMARY:
This study is designed to look at the effectiveness of a new technology call Nanotechnology Biomarker Tagging (NBT) in detecting COVID-19 infection using breath samples of patients. Participation in this study is expected to take less than one month and will consist of a breath sample being taken by the research team, a cheek swab being taken by the research team, a questionnaire that will be completed by the participant with the help of the research teams, and a review of your medical record.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Patients that present for COVID-19 testing, have tested Covid negative, or Covid Positive patients.

Exclusion Criteria:

* Unable to consent
* Patients on a ventilator
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of particpants who are receiving Covid-19 testing, as well as in-patient and out-patients with Covid-19.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Provide an adequate sample and compare the signals given from the two groups. | 10 minutes
  The samples from the participants will be analyzed to identify the different signals given from Covid-19 positive patients and Covid-19 negative patients

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No